CLINICAL TRIAL: NCT00908726
Title: Population Pharmacokinetic and Pharmacodynamic Modeling of Microemulsion Propofol in Healthy Volunteers: Comparison With Lipid Emulsion Propofol
Brief Title: Population Pharmacokinetics/Pharmacodynamics (PK/PD) of Microemulsion Propofol in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Gyu-Jeong Noh, Professor of department of anesthesiology and pain medicine, and Clinical pharamcology, Asan Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Microemulsion Phase 1
Record Dates: First submitted 2009-05-22; First posted 2009-05-27 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Microemulsion propofol (Experimental)
  Interventions: Drug: propofol
- Lipid emulsion propofol (Active Comparator)
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — Each subject received both propofol formulations in a crossover fashion separated by a 7-day washout period, and the order of the drug administration was randomized. Subjects received both propofol formulations (Lipid emulsion propofol: Diprivan® and Microemulsion propofol: AquafolTM) during 60 min. The infusion rate was assigned according to a nonblinded, randomized design to 1.5, 3, 6, or 12 mg/kg/hr.
  Other Names: Microemulsion propofol: AquafolTM; Lipid emulsion propofol: Diprivan®

SUMMARY:
AquafolTM (Daewon Pharmaceutical Co., Ltd., Seoul, Korea) is a microemulsion propofol that has been developed for eliminating lipid solvent-related adverse events of long chain triglyceride emulsion (LCT) propofol (Diprivan®; AstraZeneca, London, United Kingdom), such as infection, fat embolism, hypertriglyceridemia and pancreatitis. Originally, AquafolTM was formulated with 8% polyethylene glycol 660 hydroxystearate (Solutol HS 15, BASF Company Ltd., Seoul, Korea) and 5% tetrahydrofurfuryl alcohol polyethylene glycol ether (Glycofurol, Roche, Basle, Switzerland). A phase 1 study to assess the safety and tolerability of polymeric vehicles of this formulation in healthy volunteers showed dose-limiting toxicity. Subsequently, it was reformulated with 10% purified poloxamer 188 (PP188) as a nonionic block copolymer surfactant and 0.7% polyethylene glycol 660 hydroxystearate as a nonionic surfactant. Alterations in propofol formulation may result in altered pharmacokinetic, pharmacodynamic characteristics.

The aim of this study was to compare the pharmacokinetics and pharmacodynamics of propofol microemulsion and lipid emulsion, using noncompartmental analysis and population analysis with mixed effects modeling.

DETAILED DESCRIPTION:
The Subjects fasted for 6 h before study drug administration. An 18-gauge angiocatheter was placed in a vein of the antecubital area. A second angiocatheter was placed in the contralateral radial artery for frequent blood sampling. Subjects were monitored with electrocardiography, pulse oximetry, end-tidal carbon dioxide concentration, and invasive blood pressure measurement (Datex-Ohmeda S/5;Planar Systems, Inc., Beaverton, OR) and Bispectral Index (BIS) (Aspect 2000; Aspect Medical Systems, Inc., Newton,MA). In addition, the electroencephalographic activity of seven monopolar channels (Fp1, Fp2, F3, F4, Cz, P3, and P4, referenced by A2) was recorded by QEEG-8 (LXE3208, Laxtha Inc., Daejeon, Korea).

The subjects were stratified into three age groups (19-40, 41-64, and > 65 yr), and each group included 10 male and 10 female volunteers. Each subject received both propofol formulations in a crossover fashion separated by a 7-day washout period, and the order of the drug administration was randomized. Subjects received both propofol formulations during 60 min. The infusion rate was assigned according to a nonblinded, randomized design to 1.5, 3, 6, or 12 mg/kg/hr.

Samples were collected in ethylenediaminetetraacetic acid (EDTA) tube and centrifuged for 10 min at 3,500rpm. Plasma was stored at -70°C until assay. Arterial blood samples (4 ml) were taken at preset intervals: 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 15, 20, 30, 40, 50, 58, 60, 62, 66, 70, 80, 90, 120 and 150 min after administration of propofol. Venous blood samples (4ml) were taken at preset intervals: 180, 240, 300, 600, 720 and 1,200 min after administration of propofol. In addition, arterial samples were drawn when LOC (loss of consciousness) and ROC (recovery of consciousness) were observed.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 or 2 (healthy or mild systemic illness) healthy volunteers
* age ≥ 19 yr

Exclusion Criteria:

* ASA 3 or above
* out with age group above
* contraindications against the use of propofol
* abnormal laboratory finding with clinical significance
* evidence of pregnancy
* history of alcohol or drug abuse
* neurological or psychiatric disease
* unable or unwilling to give informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The aim of this study was to compare the pharmacokinetics and pharmacodynamics of microemulsion and lipid emulsion propofol. | Between 5/2/2009 until 5/31/2010

CONTACTS AND LOCATIONS:
Overall Officials: Gyu-Jeong Noh, M.D. & Ph.D., Study Chair — Professor & Chairperson, Department of Clinical Pharmacology and Therapeutics, Asan Medical Center; Byung-Moon Choi, M.D., Principal Investigator — Staff Anesthesiologist, Department of Anesthesiology and Pain Medicine, National Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Kim KM, Choi BM, Park SW, Lee SH, Christensen LV, Zhou J, Yoo BH, Shin HW, Bae KS, Kern SE, Kang SH, Noh GJ. Pharmacokinetics and pharmacodynamics of propofol microemulsion and lipid emulsion after an intravenous bolus and variable rate infusion. Anesthesiology. 2007 May;106(5):924-34. doi: 10.1097/01.anes.0000265151.78943.af. PMID 17457123
- [Background] Lee EH, Lee SH, Park DY, Ki KH, Lee EK, Lee DH, Noh GJ. Physicochemical properties, pharmacokinetics, and pharmacodynamics of a reformulated microemulsion propofol in rats. Anesthesiology. 2008 Sep;109(3):436-47. doi: 10.1097/ALN.0b013e318182a486. PMID 18719441